CLINICAL TRIAL: NCT02718729
Title: Anastomotic Leakage Following Laparoscopic Resection for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Mostafa shalaby, MD, MSc, PhD, Dr, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MD 84
Record Dates: First submitted 2016-03-12; First posted 2016-03-24 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Anastomotic Leakage
Keywords: Anastomotic leakage; Rectal cancer; Laparoscopic; Rectal resection
MeSH Terms: conditions — Anastomotic Leak; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rectal cancer patients (Other): All patients who will fulfill the inclusions criteria. Patients will undergo formal curative radical Laparoscopic resection for rectal cancer
  Interventions: Procedure: Laparoscopic resection for rectal cancer

INTERVENTIONS:
Procedure: Laparoscopic resection for rectal cancer — Formal curative radical laparoscopic rectal resection.

SUMMARY:
Anastomotic leak (AL) is a breakdown of a suture line in a surgical anastomosis with a subsequent leakage of the luminal content. Anastomotic leakage occurs commonly in rectal and esophageal anastomosis than the other parts of the alimentary tract due to technical difficulties in accessing these areas and their easily compromised blood supply.

Anastomotic leakage is the most feared complication following rectal resection and anastomosis. The incidence of anastomotic leakage ranges from 2.8% to more than 15%, with mortality rate more than 30%. Subclinical anastomotic failure may occur in up to 51% of patients.

Anastomotic leakage leads to increase the rate of secondary interventions, re-operations, longer postoperative hospital stay, increased cost, and major impact on the patient's quality of life. In the medium to long term, patient may be unfit for post-operative adjuvant therapy with decreased the disease survival. Furthermore anastomotic leakage itself may increase the local recurrence, a reduction in overall survival, and a large proportion of patients are left with a permanent stoma.

DETAILED DESCRIPTION:
Study populations: all patients will sign an informed consent prior to the surgery to be included in the study, after explanation of the nature of the disease, possible treatment, and the possibility of stoma formation.

Data recording: basic demographic data are recorded including age and sex of the patient as well as detailed information on history, risk factors, preoperative diagnostics, surgical procedure, intraoperative findings, histopathological work-up, and postoperative course.

Variables analysis: the variables are divided into patient-related, tumor-related, therapy-related, and techniques-related variables.

Preoperative workup: all patients will have detailed clinical history and physical examination including DRE. Routine laboratory investigations also are included e.g. CBC, blood glucose level, liver, and kidney function tests.

Regular workup for rectal cancer are included; full colonoscopy with biopsy, gastrografin/barium enema, TRUS evaluate degree of invasion of the rectal wall and regional lymph nodes, abdominal and pelvic CT scan, Chest x-ray or CT scan, CEA level, and EORTC Quality of life Questionnaire.

Level of the tumor: is measured from the lower border of the tumor to the anal verge by the rigid sigmoidoscope; considering it low < 6 cm, middle 6-12 cm, and upper > 12 cm.

Preoperative preparation: all patients will have preoperative mechanical bowel preparation and adequate thromboembolic prophylaxis. Prophylactic antibiotics will be given 30 - 60 minutes before surgery. A surgeon or stoma therapist will mark the site of the stoma before the operation in all patients.

Level of the anastomosis: is measured from the anastomosis to the anal verge by the rigid sigmoidoscope intraoperative; considering it low < 10 cm, middle 10-15 cm, and upper > 15 cm.

The rectal anastomosis is tested intraoperative with: trans-anal air insufflation with the pelvis immersed with saline to detect bubbles, trans-anal introduction of dye, or competence of donuts in stapled anastomosis.

Postoperative follow up:

Access the postoperative condition locally and systemically by bedsides clinical parameters, and usual blood tests like leucocyte count and CRP level at the 3rd and the 7th day postoperative.

Radiological follow up by Gastrografin enema around the 10th day or before dismissal from the hospital. Abdominal and pelvic CT scan is ordered in patients with clinical deterioration, abnormal abdominal findings, and turbid drainage secretion.

Peritoneal samples are collected from the abdominal drains at the first, third, and fifth days postoperatively for peritoneal microbiological study and cytokines (IL-6, IL-10, and TNF) level measurement.

Patients will receive a Quality of Life questionnaire (EORTC 30, 38) preoperatively, 30 days postoperative, and 30 days after stoma closure in case of diversion.

Follow up of patients continue till discharge, and 30 days postoperative. In cases with diversion follow up will continue till closure of stoma and 30 days after closure. Stoma closure in an uneventful course will be scheduled 8-10 weeks after the primary operation.

Diagnosis of leakage:

1. Fecal secretion via indwelling abdominal drainage, surgical wound or vagina.
2. Radiological via fluid collection adjacent to anastomosis associated with extraluminal contrast extravasation.

Classification of leakage: patients classified according to leakage into:

1. Non leakage group.
2. Leakage group, radiological is asymptomatic and detected on imaging, localized is diagnosed on radiological findings of a pelvic collection and clinically do not require a laparotomy or laparoscopy, and generalized is confirmed at laparotomy or laparoscopy.

Outcomes:

Primary outcomes:

Incidences of anastomotic leakage following laparoscopic resection for rectal cancer.

30 day's postoperative morbidity and mortality. secondary outcomes: The role of diversion on prevention of anastomotic leakage, are patients with diversion have low incidences of leakage.

Management of anastomotic leakage. Effect of anastomotic leakage on oncological outcome, assessment of local recurrence after 24 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo laparoscopic resection for biopsy proven rectal cancer.

Exclusion Criteria:

* Open surgery,
* Emergency intervention,
* Palliative resection,
* Stage IV with distant metastasis,
* Recurrent cancer,
* Multivisceral resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of anastomotic leakage | 2 years
  Incidence of anastomotic leakage in patients who underwent laparoscopic resection of rectal cancer. This including clinical and sub-clinical (radiological diagnosis) leakage.

SECONDARY OUTCOMES:
Role of diversion in prevention of anastomotic leakage. | 2 years
  Do the patients with diversion have low incidences of anastomotic leakage compared to those without.
Management of anastomotic leakage | 2 years
  The comparison of conservative, radio-logical, or surgical options.
Oncological outcomes of anastomotic leakage | 2 years
  For patients who complete 24 months of follow-up for local recurrence.
30 days postoperative morbidity and mortality | 30 days
  In the first 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Shalaby, M,D., MSc., Principal Investigator — Mansoura University/ University of Rome Tor Vergata
Locations (2):
- Mansoura University Hospitals, Al Mansurah, Al Dakhlia, Egypt
- Policlinico Tor Vergata Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided